CLINICAL TRIAL: NCT05720195
Title: Assessment of Prognostic Accuracy of Albumin-Bilirubin and Platelet-Albumin-Bilirubin Grades in Hepatocellular Carcinoma Patients According to Different Treatment Modalities
Brief Title: ALBI and PALBI Scores and HCC Prognosis
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Abudeif Abdelaal, MD, Principal investigator, Sohag University
Other Study IDs: Soh-Med-21-10-41
Record Dates: First submitted 2023-01-19; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Hepatocellular Carcinoma (HCC) Prognosis
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ALBI — Albumin-Bilirubin and Platelet-Albumin-Bilirubin Grades for prognosis of HCC
  Other Names: PALBI

SUMMARY:
To compare the predictive ability of ALBI and PALBI grades with CTP and MELD scores.

To investigate the efficacy of ALBI and PALBI grades for predicting the prognosis of HCC and overall survival among different modalities of treatment.

ELIGIBILITY:
Inclusion Criteria:

• The diagnosis of HCC will be based on the presence of an arterial hypervascular focal lesion > 2 cm with rapid wash-out with a single imaging modality (triphasic computed tomography (CT), or dynamic magnetic resonance imaging (MRI)) or two imaging modalities demonstrating the before mentioned feature for lesions < 2 cm with or without elevated serum alpha-fetoprotein (AFP) levels.

Exclusion Criteria:

* Patients below 18 years old.
* Patients with pre-existing other malignancies.
* Patients with pre-existing gall bladder stones, benign strictures, or other biliary diseases.
* Patients with pre-existing haematologic disorders.
* Patients with proteinuria.
* Missed follow-up.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include all patients diagnosed with HCC both males and females equal to or above 18 years old, attending the outpatient clinic or admitted at the inpatient section of Tropical Medicine and Gastroenterology Department, Sohag University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 645 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival among HCC patients as assessed by the albumin-bilirubin (ALBI) score | 2 years
  We will compare the ability of ALBI score to predict overall survival among HCC patients versus Child Pugh and MELD scores
Overall survival among HCC patients as assessed by the platelet-albumin-bilirubin (PALBI) score | 2 years
  We will compare the ability of PALBI score to predict overall survival among HCC patients versus Child Pugh and MELD scores

SECONDARY OUTCOMES:
Overall survival among HCC patients according to treatment modality as assessed by the albumin-bilirubin (ALBI) score | 2 years
  We will compare the ability of ALBI score to predict overall survival among HCC patients stratified according to treatment modality (Surgical resection, local ablation, trans-arterial chemoembolization, sorafenib and best supportive care)
Overall survival among HCC patients according to treatment modality as assessed by the platelet-albumin-bilirubin (PALBI) | 2 years
  We will compare the ability of PALBI score to predict overall survival among HCC patients stratified according to treatment modality (Surgical resection, local ablation, trans-arterial chemoembolization, sorafenib and best supportive care)

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No